CLINICAL TRIAL: NCT05417568
Title: Oxalate-Driven Host Responses in Kidney Stone Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tanecia Mitchell, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB-300009093; R01DK129885 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stones
Keywords: Kidney stones; Dietary oxalate
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Experimental): Healthy participants will randomly receive either high (250mg) or low (40mg) oxalate diet for for four days, a ten day "washout" period on a self-selected diet, and finally the opposite diet from the first for the last four days.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: High Oxalate Diet
- Calcium Oxalate Kidney Stone (Experimental): Calcium oxalate kidney stone participants will randomly receive either high (250mg) or low (40mg) oxalate diet for for four days, a ten day "washout" period on a self-selected diet, and finally the opposite diet from the first for the last four days.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: High Oxalate Diet

INTERVENTIONS:
Dietary Supplement: Low Oxalate Diet — Participants will consume a diet that is controlled in its daily contents of oxalate and calcium, and in its content of carbohydrate, fat, and protein. Participants will be asked not to take any dietary supplements, exercise strenuously, or consume food or drink that is not provided to them.
Dietary Supplement: High Oxalate Diet — Participants will consume a diet that is controlled in its daily contents of oxalate and calcium, and in its content of carbohydrate, fat, and protein. Participants will be asked not to take any dietary supplements, exercise strenuously, or consume food or drink that is not provided to them.

SUMMARY:
This study is looking to understand the role of oxalate on kidney stone development and immunity. This study will enroll healthy participants and participants with calcium oxalate kidney stones (CaOx KS). Participants will be in this study for about 3 weeks, consume controlled diets, and provide blood and urine specimens.

DETAILED DESCRIPTION:
The purpose of this longitudinal study is to examine the effects of dietary oxalate on nanocrystalluria and the immune system. Oxalate is a small molecule found in plants and plant-derived food. It has been shown that meals containing high amounts of oxalate can increase urinary oxalate excretion, which is a risk factor for calcium oxalate kidney stones (CaOx KS). Small increases in oxalate can stimulate urinary crystals to form which can elicit an immune response. This study consists of having healthy subjects and patients with CaOx KS consume both low and oxalate enriched diets to evaluate the effect of oxalate on urinary crystals and immune responses. Participants will receive a low or high oxalate diet for 4 days prior to having a wash-out period for 6 days. Participants will then crossover to the opposite oxalate diet for four more days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 60 years old.
* Able to provide informed consent.
* BMI between 20-30 kg/m2.
* Non-tobacco users or not pregnant/breastfeeding/nursing.
* Normal fasting blood comprehensive metabolic panel, complete blood count, C-reactive protein, and urinalysis. Must accurately collect two 24-hour urine collections within 20% of the appropriate ratio of creatinine (mg)/body weight (kg) for respective gender.
* Healthy subjects: No history of CaOx KS or other medical conditions.
* Patients with CaOx KS: Recent stone composition > 50% CaOx; no uric acid, struvite, or carbonate apatite stone content. Must be first-time or recurrent CaOx stone former (last stone event ≤ 3 years).
* Willing to not consume supplements (i.e. vitamins, Ca (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, and probiotics) for 2 weeks before the study and during the study.
* Willing to abstain from vigorous exercise during the study as this may compromise immune function.
* Willing to consume diets provided only by the UAB CCTS Bionutrition Core. No food allergies or intolerance to any of the foods on the study menus.
* Willing to accurately collect 24-hour urine samples, and to have blood drawn throughout the study.
* If on medications for KS prevention (e.g. thiazides, citrate supplementation excluding calcium citrate), patients must be on a stable dose regimen for at least 8 weeks prior to and during screening, with no changes in dosing anticipated during the study. Patients should not take allopurinol for 2 weeks prior to screening since allopurinol has antioxidant properties.

Exclusion Criteria:

* Failure to meet the inclusion criteria or physician refusal.
* Inability to sign and read the informed consent.
* Any medical, psychiatric, or social conditions that would prohibit participants from abiding by the study requirements.
* BMI ˃30 kg/m2 and <20 kg/m2
* Tobacco users or pregnant or breastfeeding/nursing women.
* Abnormal fasting blood comprehensive metabolic panel, complete blood count, C-reactive protein, and urinalysis. Inaccurate 24-hour urine collections.
* Healthy subjects: Currently taking or have recently taken medications within the last 3 months (i.e. antibiotics) or dietary supplements. History of KS or any medical condition that could influence absorption or excretion of oxalate.
* Active illness including COVID-19, flu, common cold, fever, diarrhea, urinary tract infections, or other infections 14 days before the study and throughout the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary Oxalate | Days 3-4 and 13-14
  Twenty-four hour urinary oxalate will be reported as mg/day.
Change in Nanocystalluria | Days 3-4 and 13-14
  Nanocrystalluria will be reported as particles/ml.
Monocyte Cellular Bioenergetics and Mitochondrial Function | Day 1
  Cellular bioenergetics and mitochondrial function will be reported as oxygen consumption rate (pmol/min/10,000 cells).
Monocyte Cellular Bioenergetics and Mitochondrial Function | Day 4
  Cellular bioenergetics and mitochondrial function will be reported as oxygen consumption rate (pmol/min/10,000 cells).
Monocyte Cellular Bioenergetics and Mitochondrial Function | Day 11
  Cellular bioenergetics and mitochondrial function will be reported as oxygen consumption rate (pmol/min/10,000 cells).
Monocyte Cellular Bioenergetics and Mitochondrial Function | Day 14
  Cellular bioenergetics and mitochondrial function will be reported as oxygen consumption rate (pmol/min/10,000 cells).
Monocyte Subtypes | Day 1
  Monocyte subtypes will be determined using flow cytometry (mean fluorescence intensity).
Monocyte Subtypes | Day 4
  Monocyte subtypes will be determined using flow cytometry (mean fluorescence intensity).
Monocyte Subtypes | Day 11
  Monocyte subtypes will be determined using flow cytometry (mean fluorescence intensity).
Monocyte Subtypes | Day 14
  Monocyte subtypes will be determined using flow cytometry (mean fluorescence intensity).
Monocyte Transcriptomics | Day 1
  Monocyte transcriptomics will be reported as gene expression (mRNA levels)
Monocyte Transcriptomics | Day 4
  Monocyte transcriptomics will be reported as gene expression (mRNA levels)
Monocyte Transcriptomics | Day 11
  Monocyte transcriptomics will be reported as gene expression (mRNA levels)
Monocyte Transcriptomics | Day 14
  Monocyte transcriptomics will be reported as gene expression (mRNA levels)

CONTACTS AND LOCATIONS:
Overall Officials: Tanecia Mitchell, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States